CLINICAL TRIAL: NCT00306748
Title: A Randomized, Multicenter, Double-Blind, Parallel-Design, Phase 2 Trial of Oral MD-1100 Acetate Administered for 14 Days Once Daily at 100 ug, 300 ug, 1000 ug, or Placebo to Patients With Chronic Constipation
Brief Title: Phase 2 Study of MD-1100 Acetate Administered for 14 Days to Patients Meeting Criteria for Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCP-103-004
Record Dates: First submitted 2006-03-20; First posted 2006-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Constipation
Keywords: Chronic Constipation; Chronic Idiopathic Constipation; Constipation; CIC; CC; MD-1100; MD-1100 Acetate; Microbia; Microbia, Inc.; linaclotide; linaclotide acetate
MeSH Terms: conditions — Constipation | interventions — linaclotide

INTERVENTIONS:
Drug: MD-1100 Acetate

SUMMARY:
The purpose of this study is to determine the safety and gastrointestinal pharmacodynamics (stool frequency, stool consistency, stool ease of passage, stool completeness of evacuation) of MD-1100 acetate administered daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breastfeeding female, age 18-70 years old at the time of first dose;
* Sexually active patients of childbearing potential agree to use double-barrier birth control;
* Females of childbearing potential must complete negative pregnancy tests prior to first dose;
* Negative colonoscopy within 10 years or completion of negative flexible sigmoidoscopy if under the age of 50 provided there is no history of rectal bleeding, weight loss, or anemia;
* BMI must be greater than/equal to 18.5 and less than 35.0;
* Successful completion of physical exam, 12-lead ECG, clinical laboratory tests prior to first dose of study medication;
* Vital signs must not have clinically-significant findings within 4 hours of first dose of study medication;
* Patient reports 3 or less spontaneous bowel movements (SBMs) per week and meets 1 or more of the following criteria for constipation for 12 weeks in the previous 12 months: straining at least 25% bowel movements (BMs), lumpy or hard stools at least 25% of BMs, or sensation of incomplete evacuation at least 25% of BMs;
* Patient reports 3 or less SBMs during the 7-day Pre-treatment Period;
* Patient is compliant with IVRS for at least 6 days in the 7-day Pre-treatment Period.

Exclusion Criteria:

* Use of investigational drug within 30 days;
* Laxative/enema-induced diarrhea within 60 days;
* Patient meets ROME II criteria for functional diarrhea;
* Most bothersome symptom is moderate or severe abdominal pain or abdominal discomfort;
* History of cancer, inflammatory bowel disease, ischemic colitis, bowel resection, colostomy, or fecal impaction;
* Diagnosis of cathartic colon or laxative/enema abuse, pelvic floor dysfunction, evacuation disorder, bulimia, anorexia, or neurological disorders;
* Surgery within 30 days or GI surgery within 6 months of first dose of study medication. Cholecystectomy and/or appendectomy are acceptable if completed more than 60 days prior to first dose of study medication;
* Patient may not use any disallowed medications (prescription and/or over-the-counter treatments for chronic constipation or C-IBS, drugs that target 5-HT4, 5-HT2b, or 5-HT3 receptors, narcotics, anti-cholinergic agents, GI preparations, etc.) during the 7-day Pre-treatment Period or during the study. Stable, continuous (30 days or more) use of dietary fiber is acceptable.
* Any acute or chronic condition that would limit the patient's ability to complete and/or participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-03; Study Completion 2006-08

PRIMARY OUTCOMES:
Safety will be evaluated on an ongoing basis by completing physical examinations, ECGs, clinical laboratory tests, and adverse event reporting.

SECONDARY OUTCOMES:
Stool Frequency will be reported daily
Stool Consistency (Bristol Stool Form Scale) will be reported daily
Stool Ease of Passage will be reported daily
Stool Completeness of Evacuation will be reported daily
Patient Assessment of Abdominal Discomfort will be reported weekly
Patient Assessment of Constipation will be reported weekly
Patient Assessment of Overall Relief will be reported weekly
Part 1 of the Irritable Bowel Symptom Severity Scale (IBSSS) will be reported once pre-dose and once post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Johnston, MD, FACP, Study Director — Microbia, Inc.
Locations (14):
- United States (14):
  - Clinical Research Associates, Huntsville, Alabama
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Consultants for Clinical Research of South Florida, Boynton Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Chung H. Kim, MD, Pittsford, New York
  - UC for Functional GI & Motility Disorders, Chapel Hill, North Carolina
  - Vital Research, Greensboro, North Carolina
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - ClinSearch, Chattanooga, Tennessee
  - Memphis Gastroenterology Clinic, Germantown, Tennessee
  - Austin Gastroenterology, P.A., Austin, Texas
  - Trinity Clinic - Corsicana, Corsicana, Texas
  - East Coast Clinical Research, LLC, Virginia Beach, Virginia
  - Vantage Clinical Research, Olympia, Washington